CLINICAL TRIAL: NCT06572748
Title: Evaluation Study for the Chef Anchor 3.0 Program for Older People With Mild Cognitive Impairment/Dementia and Their Informal Caregivers
Brief Title: Evaluation Study for the Chef Anchor 3.0 Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Hong Kong Sheng Kung Hui Welfare Council Limited (Other)
Responsible Party: Principal Investigator, Dr. Pui-Hing Chau, Associate Professor, The University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EA240323
Record Dates: First submitted 2024-08-20; First posted 2024-08-27 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Mild Cognitive Impairment; Dementia
MeSH Terms: conditions — Cognitive Dysfunction; Dementia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assigned intervention (Other): During the first 10 weeks, the intervention group will undergo the 10-week programme in the "Chef Anchor 3.0"
  Interventions: Other: 10-week programme
- Assigned waitlist attention control (Other): During the first 10 weeks, no activity for the waitlist control group. Then, from week 10 to 20, the waitlist control group will attend the same 10-week programme.
  Interventions: Other: 10-week programme

INTERVENTIONS:
Other: 10-week programme — 1. 2-week health education (4 sessions, 60 minutes per session) Social workers and occupational therapists will explain the cognitive training elements of the program and introduce the "DementiAbility Methods" to the participants. Nutritionist, speech therapists, and Chinese medicine practitioner will share insights from their perspectives to enhance participants' understanding of cognitive impairments.
  2. 8-week cooking class (5 sessions, 120 minutes per session) The culinary instructor will teach participants to cook homemade dishes while integrating "procedural memory" into recipes. Older adults and their caregivers will cook together based on the "procedural recipe" designed by caregivers, aiming to enhance communication between them and create joyful memories. The cooking class will begin with 20-30 minutes an interactive nutrition-based session. The session themes will focus on healthy diet and food safety. Participants will be able to ask questions and make comments.

SUMMARY:
Objectives:

1. (Primary)To estimate the potential effects of the cooking program on the people with MCI/dementia and their informal caregivers;
2. To investigate if the potential effects can be maintained after the completion of the program.

Study design and participants:

A convenience sample of 68 pair older adults with MCI/dementia and their informal caregivers from the Chef Anchor 3.0 Programme will be referred to the research team. Overall, participants will be assigned to intervention group and waitlist control group in a ratio of 1:1. Allocation will take into account the participants' availability and the programme capacity. Assessors of outcomes and data analyst will be blinded throughout the whole study.

During the first 10 weeks, the intervention group will undergo the 10-week programme in the "Chef Anchor 3.0", while no activity for the waitlist control group. Then, from week 10 to 20, the waitlist control group will attend the same 10-week programme.

Measurements:

Main outcome measures for people with MCI/dementia will include confidence in cooking (Primary), cooking capability, satisfaction with autonomy in cooking, Satisfaction with meal choices, Worried about future cooking ability and meal choices, cognitive function, self-reported appetite, psychological well-being, family harmony and satisfaction, as well as self-rated health.

Outcome measures for informal caregivers will include confidence in care recipient' s cooking, worried about future cooking ability and meal choices of care recipient, caregiver burden, psychological well-being, family harmony and satisfaction, as well as self-rated health.

Other measures will include attendance rate, home practice rate, drop-out rate, programme satisfaction, and recommendation to others.

Hypotheses

1. The confidence in cooking, cooking capability, satisfaction with autonomy in cooking, satisfaction with meal choices, worried about future cooking ability and meal choices, cognitive function, self-reported appetite, psychological well-being, family satisfaction, and self-rated health of older adults with MCI/dementia would improve after the programme;
2. The confidence in care recipient's cooking, worried about future cooking ability and meal choices of care recipient, psychological well-being, family satisfaction, caregiver burden, and self-rated health of informal caregivers would improve after the programme;
3. The 10-week programme is acceptable for the most of older adults with MCI/dementia and their informal caregivers.

ELIGIBILITY:
Inclusion Criteria:

i. Aged 60 or above;

ii. Diagnosed by medical doctor has having MCI/dementia as reported by the older adults or their informal caregivers, or with reported subjective decline of cognitive function and with 5-min MoCA score ≤7th age- and education-specific percentile (Wong et al., 2015);

iii. Ability to follow simple instructions;

iv. Adequate physical strength to attend cooking workshops.

Exclusion Criteria:

i. Without caregiver

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline confidence in cooking of people with MCI/dementia at 10 weeks | 10 weeks after baseline
  measured by a single question asking to what extent (1 to 10) the participant feels confident with cooking a meal. Score 1 refers to no confidence and score 10 refers to very confident. Ten smileys will be used to visualize the different extent. This outcome is the primary outcome.
Change from baseline confidence in cooking of people with MCI/dementia at 20 weeks | 20 weeks after baseline
  measured by a single question asking to what extent (1 to 10) the participant feels confident with cooking a meal. Score 1 refers to no confidence and score 10 refers to very confident. Ten smileys will be used to visualize the different extent. This outcome is the primary outcome.
Change from baseline confidence in cooking of people with MCI/dementia at 30 weeks | 30 weeks after baseline, only for waitlist control group
  measured by a single question asking to what extent (1 to 10) the participant feels confident with cooking a meal. Score 1 refers to no confidence and score 10 refers to very confident. Ten smileys will be used to visualize the different extent. This outcome is the primary outcome.

SECONDARY OUTCOMES:
Change from baseline cooking capability of people with MCI/dementia at 10 weeks | 10 weeks after baseline
  measured by a single question asking how much assistance from others the participant is needed when cooking. Score 0 refers to never cook, score 1 refers to being able to cook independently, score 2 refers to sometimes or part of the process requires help from others or requiring special assistive equipment/devices, and score 3 refers to being dependent on help from others or unable to complete this activity due to health condition.
Change from baseline cooking capability of people with MCI/dementia at 20 weeks | 20 weeks after baseline
  measured by a single question asking how much assistance from others the participant is needed when cooking. Score 0 refers to never cook, score 1 refers to being able to cook independently, score 2 refers to sometimes or part of the process requires help from others or requiring special assistive equipment/devices, and score 3 refers to being dependent on help from others or unable to complete this activity due to health condition
Change from baseline cooking capability of people with MCI/dementia at 30 weeks | 30 weeks after baseline, only for waitlist control group
  measured by a single question asking how much assistance from others the participant is needed when cooking. Score 0 refers to never cook, score 1 refers to being able to cook independently, score 2 refers to sometimes or part of the process requires help from others or requiring special assistive equipment/devices, and score 3 refers to being dependent on help from others or unable to complete this activity due to health condition.
Change from baseline satisfaction with autonomy in cooking of people with MCI/dementia at 10 weeks | 10 weeks after baseline
  measured by a single question asking to what extent (1 to 10) the participant is satisfied with the ability to cook a meal autonomously. Score 1 refers to not satisfactory at all and score 10 refers to very satisfactory. Ten smileys will be used to visualize the different extent.
Change from baseline satisfaction with autonomy in cooking of people with MCI/dementia at 20 weeks | 20 weeks after baseline
  measured by a single question asking to what extent (1 to 10) the participant is satisfied with the ability to cook a meal autonomously. Score 1 refers to not satisfactory at all and score 10 refers to very satisfactory. Ten smileys will be used to visualize the different extent.
Change from baseline satisfaction with autonomy in cooking of people with MCI/dementia at 30 weeks | 30 weeks after baseline, only for waitlist control group
  measured by a single question asking to what extent (1 to 10) the participant is satisfied with the ability to cook a meal autonomously. Score 1 refers to not satisfactory at all and score 10 refers to very satisfactory. Ten smileys will be used to visualize the different extent.
Change from baseline satisfaction with meal choices of people with MCI/dementia at 10 weeks | 10 weeks after baseline
  measured by two questions asking to what extent (1 to 10) the participant is satisfied with the choice of ingredients and cooking methods, respectively. Score 1 refers to not satisfactory at all and score 10 refers to very satisfactory. Ten smileys will be used to visualize the different extent.
Change from baseline satisfaction with meal choices of people with MCI/dementia at 20 weeks | 20 weeks after baseline
  measured by two questions asking to what extent (1 to 10) the participant is satisfied with the choice of ingredients and cooking methods, respectively. Score 1 refers to not satisfactory at all and score 10 refers to very satisfactory. Ten smileys will be used to visualize the different extent.
Change from baseline satisfaction with meal choices of people with MCI/dementia at 30 weeks | 30 weeks after baseline, only for waitlist control group
  measured by two questions asking to what extent (1 to 10) the participant is satisfied with the choice of ingredients and cooking methods, respectively. Score 1 refers to not satisfactory at all and score 10 refers to very satisfactory. Ten smileys will be used to visualize the different extent.
Change from baseline worried about future cooking ability and meal choices of people with MCI/dementia at 10 weeks | 10 weeks after baseline
  measured by three questions to what extent (1 to 10) the participant is worried about with the future cooking ability, choice of ingredients and cooking methods, respectively. Score 1 refers to completely worried and score 10 refers to not worried at all. Ten smileys will be used to visualize the different extent.
Change from baseline worried about future cooking ability and meal choices of people with MCI/dementia at 20 weeks | 20 weeks after baseline
  measured by three questions to what extent (1 to 10) the participant is worried about with the future cooking ability, choice of ingredients and cooking methods, respectively. Score 1 refers to completely worried and score 10 refers to not worried at all. Ten smileys will be used to visualize the different extent.
Change from baseline worried about future cooking ability and meal choices of people with MCI/dementia at 30 weeks | 30 weeks after baseline, only for waitlist control group
  measured by three questions to what extent (1 to 10) the participant is worried about with the future cooking ability, choice of ingredients and cooking methods, respectively. Score 1 refers to completely worried and score 10 refers to not worried at all. Ten smileys will be used to visualize the different extent.
Change from baseline cognitive function of people with MCI/dementia at 10 weeks | 10 weeks after baseline
  measured by the Chinese version of 5-min Montreal Cognitive Assessment (MoCA) (Feng et al., 2021; A. Wong et al., 2015). The assessment comprises four parts, including memory, language fluency, orientation, and delayed recall. The total score ranged between 0 to 30, and is obtained by summing the sub-scores from each part, with a higher score indicating better cognitive function. To determine the cognitive performance of participants, their scores will be compared to their age- and education-specific standards.
Change from baseline cognitive function of people with MCI/dementia at 20 weeks | 20 weeks after baseline
  measured by the Chinese version of 5-min Montreal Cognitive Assessment (MoCA) (Feng et al., 2021; A. Wong et al., 2015). The assessment comprises four parts, including memory, language fluency, orientation, and delayed recall. The total score ranged between 0 to 30, and is obtained by summing the sub-scores from each part, with a higher score indicating better cognitive function. To determine the cognitive performance of participants, their scores will be compared to their age- and education-specific standards.
Change from baseline cognitive function of people with MCI/dementia at 30 weeks | 30 weeks after baseline, only for waitlist control group
  measured by the Chinese version of 5-min Montreal Cognitive Assessment (MoCA) (Feng et al., 2021; A. Wong et al., 2015). The assessment comprises four parts, including memory, language fluency, orientation, and delayed recall. The total score ranged between 0 to 30, and is obtained by summing the sub-scores from each part, with a higher score indicating better cognitive function. To determine the cognitive performance of participants, their scores will be compared to their age- and education-specific standards.
Change from baseline self-reported appetite of people with MCI/dementia at 10 weeks | 10 weeks after baseline
  measured by a single question asking to what extent (1 to 10) the participant agrees the appetite is good. Score 1 refers to not agree at all and score 10 refers to totally agree. Higher score indicates better appetite. Ten smileys will be used to visualize the different extent.
Change from baseline self-reported appetite of people with MCI/dementia at 20 weeks | 20 weeks after baseline
  measured by a single question asking to what extent (1 to 10) the participant agrees the appetite is good. Score 1 refers to not agree at all and score 10 refers to totally agree. Higher score indicates better appetite. Ten smileys will be used to visualize the different extent.
Change from baseline self-reported appetite of people with MCI/dementia at 30 weeks | 30 weeks after baseline, only for waitlist control group
  measured by a single question asking to what extent (1 to 10) the participant agrees the appetite is good. Score 1 refers to not agree at all and score 10 refers to totally agree. Higher score indicates better appetite. Ten smileys will be used to visualize the different extent
Change from baseline meaning in life of psychological well-being of people with MCI/dementia at 10 weeks | 10 weeks after baseline
  Measured by two questions asking to what extent (1 to 10) the participant agrees with there is purpose and meaning in life, respectively. Score 1 refers to not agree at all and score 10 refers to totally agree. Ten smileys will be used to visualize the different extent.
Change from baseline meaning in life of psychological well-being of people with MCI/dementia at 20 weeks | 20 weeks after baseline
  Measured by two questions asking to what extent (1 to 10) the participant agrees with there is purpose and meaning in life, respectively. Score 1 refers to not agree at all and score 10 refers to totally agree. Ten smileys will be used to visualize the different extent.
Change from baseline meaning in life of psychological well-being of people with MCI/dementia at 30 weeks | 30 weeks after baseline, only for waitlist control group
  Measured by two questions asking to what extent (1 to 10) the participant agrees with there is purpose and meaning in life, respectively. Score 1 refers to not agree at all and score 10 refers to totally agree. Ten smileys will be used to visualize the different extent.
Change from baseline Happiness of psychological well-being of people with MCI/dementia at 10 weeks | 10 weeks after baseline
  Measured by a single question asking about the extent of happiness in the past two months. Score 1 refers to not happy at all and score 10 refers to total happiness. Ten smileys will be used to visualize the different extent.
Change from baseline Happiness of psychological well-being of people with MCI/dementia at 20 weeks | 20 weeks after baseline
  Measured by a single question asking about the extent of happiness in the past two months. Score 1 refers to not happy at all and score 10 refers to total happiness. Ten smileys will be used to visualize the different extent.
Change from baseline Happiness of psychological well-being of people with MCI/dementia at 30 weeks | 30 weeks after baseline, only for waitlist control group
  Measured by a single question asking about the extent of happiness in the past two months. Score 1 refers to not happy at all and score 10 refers to total happiness. Ten smileys will be used to visualize the different extent.
Change from baseline food-related life satisfaction of psychological well-being of people with MCI/dementia at 10 weeks | 10 weeks after baseline
  Measured by the Satisfaction With Food-Related Life (SWFL) scale (Grunert et al., 2007). Total score ranges from 5 to 30. A higher score indicates a greater level of food-related life satisfaction.
Change from baseline food-related life satisfaction of psychological well-being of people with MCI/dementia at 20 weeks | 20 weeks after baseline
  Measured by the Satisfaction With Food-Related Life (SWFL) scale (Grunert et al., 2007). Total score ranges from 5 to 30. A higher score indicates a greater level of food-related life satisfaction.
Change from baseline food-related life satisfaction of psychological well-being of people with MCI/dementia at 30 weeks | 30 weeks after baseline, only for waitlist control group
  Measured by the Satisfaction With Food-Related Life (SWFL) scale (Grunert et al., 2007). Total score ranges from 5 to 30. A higher score indicates a greater level of food-related life satisfaction.
Change from baseline self-esteem of psychological well-being of people with MCI/dementia at 10 weeks | 10 weeks after baseline
  Measured by the Chinese version of the Rosenberg Self-Esteem Scale (RSE), containing 10 items. Higher total score indicating higher self-esteem (Yeung, 1998).
Change from baseline self-esteem of psychological well-being of people with MCI/dementia at 20 weeks | 20 weeks after baseline
  Measured by the Chinese version of the Rosenberg Self-Esteem Scale (RSE), containing 10 items. Higher total score indicating higher self-esteem (Yeung, 1998).
Change from baseline self-esteem of psychological well-being of people with MCI/dementia at 30 weeks | 30 weeks after baseline, only for waitlist control group
  Measured by the Chinese version of the Rosenberg Self-Esteem Scale (RSE), containing 10 items. Higher total score indicating higher self-esteem (Yeung, 1998).
Change from baseline family harmony and satisfaction of people with MCI/dementia at 10 weeks | 10 weeks after baseline
  measured by Chinese version of 5-item Family Harmony Scale (FHS-5) (Kavikondala et al., 2016). Five related questions asking to what extent (1 to 5) the participant agrees with the statement. These questions include (1) my family functions well for all members, (2) my family's day-to-day interactions are peaceful, (3) family members accommodate each other, (4) I am proud of my family, and (5) my family is harmonious. Score 1 refers to strongly agree, score 2 refers to agree, score 3 refers to neutral, score 4 refers to disagree, and score 5 refers to strongly disagree. Total score ranges from 5 to 25. Higher score indicates worse family harmony and satisfaction.
Change from baseline family harmony and satisfaction of people with MCI/dementia at 20 weeks | 20 weeks after baseline
  measured by Chinese version of 5-item Family Harmony Scale (FHS-5) (Kavikondala et al., 2016). Five related questions asking to what extent (1 to 5) the participant agrees with the statement. These questions include (1) my family functions well for all members, (2) my family's day-to-day interactions are peaceful, (3) family members accommodate each other, (4) I am proud of my family, and (5) my family is harmonious. Score 1 refers to strongly agree, score 2 refers to agree, score 3 refers to neutral, score 4 refers to disagree, and score 5 refers to strongly disagree. Total score ranges from 5 to 25. Higher score indicates worse family harmony and satisfaction.
Change from baseline family harmony and satisfaction of people with MCI/dementia at 30 weeks | 30 weeks after baseline, only for waitlist control group
  measured by Chinese version of 5-item Family Harmony Scale (FHS-5) (Kavikondala et al., 2016). Five related questions asking to what extent (1 to 5) the participant agrees with the statement. These questions include (1) my family functions well for all members, (2) my family's day-to-day interactions are peaceful, (3) family members accommodate each other, (4) I am proud of my family, and (5) my family is harmonious. Score 1 refers to strongly agree, score 2 refers to agree, score 3 refers to neutral, score 4 refers to disagree, and score 5 refers to strongly disagree. Total score ranges from 5 to 25. Higher score indicates worse family harmony and satisfaction.
Change from baseline self-rated health of people with MCI/dementia at 10 weeks | 10 weeks after baseline
  measured by a single question asking the participant to rate his or her health (Lam et al., 1998). Score 1 refers to excellent, score 2 refers to very good, score 3 refers to good, score 4 refers to fair, and score 5 refers to poor.
Change from baseline self-rated health of people with MCI/dementia at 20 weeks | 20 weeks after baseline
  measured by a single question asking the participant to rate his or her health (Lam et al., 1998). Score 1 refers to excellent, score 2 refers to very good, score 3 refers to good, score 4 refers to fair, and score 5 refers to poor.
Change from baseline self-rated health of people with MCI/dementia at 30 weeks | 30 weeks after baseline, only for waitlist control group
  measured by a single question asking the participant to rate his or her health (Lam et al., 1998). Score 1 refers to excellent, score 2 refers to very good, score 3 refers to good, score 4 refers to fair, and score 5 refers to poor.
Change from baseline confidence in care recipient's cooking of caregivers at 10 weeks | 10 weeks after baseline
  measured by a single question in the questionnaire asking to what extent (1 to 10) the caregiver trusts the care recipient to cook themselves. Score 1 refers to not trust at all and score 10 refers to complete trust.
Change from baseline confidence in care recipient's cooking of caregivers at 20 weeks | 20 weeks after baseline
  measured by a single question in the questionnaire asking to what extent (1 to 10) the caregiver trusts the care recipient to cook themselves. Score 1 refers to not trust at all and score 10 refers to complete trust.
Change from baseline confidence in care recipient's cooking of caregivers at 30 weeks | 30 weeks after baseline, only for waitlist control group
  measured by a single question in the questionnaire asking to what extent (1 to 10) the caregiver trusts the care recipient to cook themselves. Score 1 refers to not trust at all and score 10 refers to complete trust.
Change from baseline worried about future cooking ability and meal choices of care recipient of caregivers at 10 weeks | 10 weeks after baseline
  measured by three questions to what extent (1 to 10) the participant is worried about with the future cooking ability, choice of ingredients and cooking methods, respectively. Score 1 refers to completely worried and score 10 refers to not worried at all.
Change from baseline worried about future cooking ability and meal choices of care recipient of caregivers at 20 weeks | 20 weeks after baseline
  measured by three questions to what extent (1 to 10) the participant is worried about with the future cooking ability, choice of ingredients and cooking methods, respectively. Score 1 refers to completely worried and score 10 refers to not worried at all.
Change from baseline worried about future cooking ability and meal choices of care recipient of caregivers at 30 weeks | 30 weeks after baseline, only for waitlist control group
  measured by three questions to what extent (1 to 10) the participant is worried about with the future cooking ability, choice of ingredients and cooking methods, respectively. Score 1 refers to completely worried and score 10 refers to not worried at all.
Change from baseline caregiver burden at 10 weeks | 10 weeks after baseline
  measured by the Zarit Burden Interview (ZBI) scale (Chan et al., 2005; Schreiner et al., 2006; Zarit et al., 1980). The ZBI consists of 22 items rated on a 5-point Likert scale that ranges from 0 (never) to 4 (nearly always) with the sum of scores ranging between 0 and 88. Higher scores indicate a greater burden. A score of 17 or more was considered a high burden.
Change from baseline caregiver burden at 20 weeks | 20 weeks after baseline
  measured by the Zarit Burden Interview (ZBI) scale (Chan et al., 2005; Schreiner et al., 2006; Zarit et al., 1980). The ZBI consists of 22 items rated on a 5-point Likert scale that ranges from 0 (never) to 4 (nearly always) with the sum of scores ranging between 0 and 88. Higher scores indicate a greater burden. A score of 17 or more was considered a high burden.
Change from baseline caregiver burden at 30 weeks | 30 weeks after baseline, only for waitlist control group
  measured by the Zarit Burden Interview (ZBI) scale (Chan et al., 2005; Schreiner et al., 2006; Zarit et al., 1980). The ZBI consists of 22 items rated on a 5-point Likert scale that ranges from 0 (never) to 4 (nearly always) with the sum of scores ranging between 0 and 88. Higher scores indicate a greater burden. A score of 17 or more was considered a high burden.
Change from baseline meaning in life of psychological well-being of caregiver at 10 weeks | 10 weeks after baseline
  Measured by the Chinese version of the Meaning in Life Questionnaire. Total score ranged between 0 to 100. A higher total score indicates a greater sense of meaning in life.
Change from baseline meaning in life of psychological well-being of caregiver at 20 weeks | 20 weeks after baseline
  Measured by the Chinese version of the Meaning in Life Questionnaire. Total score ranged between 0 to 100. A higher total score indicates a greater sense of meaning in life.
Change from baseline meaning in life of psychological well-being of caregiver at 30 weeks | 30 weeks after baseline, only for waitlist control group
  Measured by the Chinese version of the Meaning in Life Questionnaire. Total score ranged between 0 to 100. A higher total score indicates a greater sense of meaning in life.
Change from baseline happiness of psychological well-being of caregiver at 10 weeks | 10 weeks after baseline
  Measured by the Chinese version of the 4-item Subjective Happiness Scale (SHS). The score is the average of the four items (1 to 7), a higher score indicates a higher level of subjective happiness.
Change from baseline happiness of psychological well-being of caregiver at 20 weeks | 20 weeks after baseline
  Measured by the Chinese version of the 4-item Subjective Happiness Scale (SHS). The score is the average of the four items (1 to 7), a higher score indicates a higher level of subjective happiness.
Change from baseline happiness of psychological well-being of caregiver at 30 weeks | 30 weeks after baseline, only for waitlist control group
  Measured by the Chinese version of the 4-item Subjective Happiness Scale (SHS). The score is the average of the four items (1 to 7), a higher score indicates a higher level of subjective happiness.
Change from baseline life satisfaction of psychological well-being of caregiver at 10 weeks | 10 weeks after baseline
  Measured by the Chinese version of the satisfaction with life scale (SWLS). Total score ranges from 5 to 35. A higher average score indicates a greater level of life satisfaction.
Change from baseline life satisfaction of psychological well-being of caregiver at 20 weeks | 20 weeks after baseline
  Measured by the Chinese version of the satisfaction with life scale (SWLS). Total score ranges from 5 to 35. A higher average score indicates a greater level of life satisfaction.
Change from baseline life satisfaction of psychological well-being of caregiver at 30 weeks | 30 weeks after baseline, only for waitlist control group
  Measured by the Chinese version of the satisfaction with life scale (SWLS). Total score ranges from 5 to 35. A higher average score indicates a greater level of life satisfaction.
Change from baseline life satisfaction of subjective well-being of caregiver at 10 weeks | 10 weeks after baseline
  Measured by the Chinese version of the World Health Organization Five Well-Being Index (WHO-5). The total raw score is multiplied by 4 to give the final score which ranges from 0 to 100, higher score indicates better well-being.
Change from baseline life satisfaction of subjective well-being of caregiver at 20 weeks | 20 weeks after baseline
  Measured by the Chinese version of the World Health Organization Five Well-Being Index (WHO-5). The total raw score is multiplied by 4 to give the final score which ranges from 0 to 100, higher score indicates better well-being.
Change from baseline life satisfaction of subjective well-being of caregiver at 30 weeks | 30 weeks after baseline, only for waitlist control group
  Measured by the Chinese version of the World Health Organization Five Well-Being Index (WHO-5). The total raw score is multiplied by 4 to give the final score which ranges from 0 to 100, higher score indicates better well-being.
Change from baseline family harmony and satisfaction of caregiver at 10 weeks | 10 weeks after baseline
  measured by Chinese version of 5-item Family Harmony Scale (FHS-5) (Kavikondala et al., 2016). Five related questions asking to what extent (1 to 5) the participant agrees with the statement. These questions include (1) my family functions well for all members, (2) my family's day-to-day interactions are peaceful, (3) family members accommodate each other, (4) I am proud of my family, and (5) my family is harmonious. Score 1 refers to strongly agree, score 2 refers to agree, score 3 refers to neutral, score 4 refers to disagree, and score 5 refers to strongly disagree. Total score ranges from 5 to 25. Higher score indicates worse family harmony and satisfaction.
Change from baseline family harmony and satisfaction of caregiver at 20 weeks | 20 weeks after baseline
  measured by Chinese version of 5-item Family Harmony Scale (FHS-5) (Kavikondala et al., 2016). Five related questions asking to what extent (1 to 5) the participant agrees with the statement. These questions include (1) my family functions well for all members, (2) my family's day-to-day interactions are peaceful, (3) family members accommodate each other, (4) I am proud of my family, and (5) my family is harmonious. Score 1 refers to strongly agree, score 2 refers to agree, score 3 refers to neutral, score 4 refers to disagree, and score 5 refers to strongly disagree. Total score ranges from 5 to 25. Higher score indicates worse family harmony and satisfaction.
Change from baseline family harmony and satisfaction of caregiver at 30 weeks | 30 weeks after baseline, only for waitlist control group
  measured by Chinese version of 5-item Family Harmony Scale (FHS-5) (Kavikondala et al., 2016). Five related questions asking to what extent (1 to 5) the participant agrees with the statement. These questions include (1) my family functions well for all members, (2) my family's day-to-day interactions are peaceful, (3) family members accommodate each other, (4) I am proud of my family, and (5) my family is harmonious. Score 1 refers to strongly agree, score 2 refers to agree, score 3 refers to neutral, score 4 refers to disagree, and score 5 refers to strongly disagree. Total score ranges from 5 to 25. Higher score indicates worse family harmony and satisfaction.
Change from baseline self-rated health of caregiver at 10 weeks | 10 weeks after baseline
  measured by a single question asking the participant to rate his or her health (Lam et al., 1998). Score 1 refers to excellent, score 2 refers to very good, score 3 refers to good, score 4 refers to fair, and score 5 refers to poor.
Change from baseline self-rated health of caregiver at 20 weeks | 20 weeks after baseline
  measured by a single question asking the participant to rate his or her health (Lam et al., 1998). Score 1 refers to excellent, score 2 refers to very good, score 3 refers to good, score 4 refers to fair, and score 5 refers to poor.
Change from baseline self-rated health of caregiver at 30 weeks | 30 weeks after baseline, only for waitlist control group
  measured by a single question asking the participant to rate his or her health (Lam et al., 1998). Score 1 refers to excellent, score 2 refers to very good, score 3 refers to good, score 4 refers to fair, and score 5 refers to poor.
Attendance rate | During 10 weeks intervention
  collected by class attendance record for face-to-face health education and cooking classes.
Home practice rate | 10, 20 weeks after baseline for intervention group. 10, 20 and 30 weeks after baseline for waitlist control group.
  collected by a single question in the questionnaire asking how many times older adults with MCI/dementia and their caregivers have practiced cooking at home in the last two months.
Drop-out rate | During 20 weeks after baseline for intervention group. During 30 weeks after baseline for waitlist control group.
  calculated by dividing the number of participants who drop-out from the study by the number of participants joining the study. If participants withdraw, reason of withdrawal will be recorded. If participants do not wish to reveal the reason of withdrawal, the project team will respect their preference.
Programme satisfaction | 20 weeks after baseline for intervention group, 30 weeks after baseline for waitlist control group.
  measured by a single question asking to what extent (1 to 10) the participant/caregiver is satisfied with the program. Score 1 refers to not satisfactory at all and score 10 refers to very satisfactory.
Recommendation to others | 20 weeks after baseline for intervention group, 30 weeks after baseline for waitlist control group.
  measured by a single question asking to what extent (1 to 10) the participant/caregiver is willing to recommend the programme to relatives or friends. Score 1 refers to not willing at all and score 10 refers to very willing to.

CONTACTS AND LOCATIONS:
Overall Officials: Pui Hing Chau, Principal Investigator — School of Nursing, The University of Hong Kong
Locations (1):
- Elderly community centre, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No